CLINICAL TRIAL: NCT04684667
Title: '' Efficacy of Propranolol in the Treatment of Infantile Hemangioma"
Brief Title: ''Efficacy of Propranolol in the Treatment of Infantile Hemangioma"
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Essam Ezzat Anees Mowannas, Principal Investigator, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Essam Mowannas
Record Dates: First submitted 2020-04-29; First posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Infantile Hemangioma
Keywords: Hemangioma; Propranolol; Beta Blockers
MeSH Terms: conditions — Hemangioma, Capillary; Hemangioma

STUDY DESIGN:
Intervention Model Description: This study will involve patients with infantile hemangiomas who will be admitted at the Assiut University Children Hospital between January 2021 and December 2021.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Propranolol Therapy (Other): This arm will involve patients with infantile hemangiomas who will be admitted at the Assiut University Children Hospital between January 2021 and December 2021.
  Interventions: Drug: Propranolol Therapy for Infantile Hemangioma

INTERVENTIONS:
Drug: Propranolol Therapy for Infantile Hemangioma — If there are no contraindications to propranolol, it will be given at initial dose of 0.5 mg /kg/day in 2-3 divided doses with feeds and the patients will be observed for clinical signs of serious adverse reactions. If the dose is tolerated, it will be maintained for four to seven days, and then it will be increased by 0.5mg/kg/day every four days to the target dose of 2mg/kg/day. The patients will be observed for 2 hours after each dose increase for the clinical signs of severe side effects.
  Other Names: Propranolol Treatment for Infantile Hemangioma

SUMMARY:
''Evaluation of the Efficacy of Propranolol in the Treatment of Infantile Hemangioma"

DETAILED DESCRIPTION:
Infantile hemangiomas (IH) are benign tumors of vascular endothelium.They are the most common tumors of infancy. They occur in about 4% of infants, though early studies were as high as 10%, probably due to the inclusion of other vascular lesions. The incidence is higher in premature infants, Caucasians, and females (by a 3 to 5:1 ratio). Advanced maternal age, multiple gestations, and placental abnormalities are also risk factors. IHs have a unique and characteristic life cycle consisting of three phases: proliferative, involuting, and involuted.

The majority of IHs do not require any specific treatment other than observation and reassurance of the parents. Even tumors that exhibit rapid growth or fiery red skin will spontaneously regress and leave behind little to no evidence of their presence. However, regular follow-up is important as the potential complications have few clinical indicators.

Reasons for treatment include dangerous locations (impinging on a vital structure such as the airway or eye), unusually large size or rapid growth, and local or endangering complications (skin ulceration or high-output heart failure). Hemangiomas exhibiting the aforementioned risk factors or complications should be considered for treatment. As hemangiomas are tumors of pure angiogenesis, pharmacologic therapy involves angiogenesis inhibition.

Historically, steroids have been used as the primary treatment for IH. Steroids have been shown to be antiangiogenic in a number of in vitro settings and also have shown good therapeutic effects clinically. However, the use of steroids may lead to various complications including gastroesophageal reflux and growth disorders, although these complications are associated with long-term use and high dose. A type of anticancer drug or immunomodulator, interferon alfa, may be used for severe IH in cases where patients did not respond to steroids. However, interferon alfa also has several possible adverse effects, including fever, muscle pain, systemic myalgia, and in severe cases, liver damage, blood toxic effects, thyroid hormonal abnormality, and neurological and neurodevelopmental toxic effects. Because of concerns about these adverse effects, many guardians of pediatric patients prefer to wait rather than accept treatment.

Propranolol, a nonselective beta blocker, has recently been recognized as an important treatment option for hemangiomas. In most centers, it has become first-line pharmacotherapy. A child with a nasal capillary hemangioma treated with propranolol for steroid-induced cardiomyopathy had regression of his lesion. This revelation led to the publication of several more studies supporting this finding. Propranolol is given orally at 2-3 mg/kg/day, in two or three divided doses, and discontinued following regression of the lesion. Treatment often leads to a consistent, rapid, therapeutic effect with softening of the lesion on palpation and color shift from intense red to purple. Propranolol is well tolerated but can cause rare side effects such as bradycardia, gastroesophageal reflux, hypoglycemia, hypotension, rash, somnolence, and wheezing.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with problematic infantile hemangiomas:

A-Large hemangiomas at increased risk of scarring or disfigurement at any site. B-Hemangiomas carrying functional risks near the eyes, nose, natural orifices, limbs, genitalia.

C-Ulcerated infantile hemangiomas. D-Uncomplicated progressive infantile hemangiomas with unpredictable future course.

E-Life-threatening hemangiomas.

* Multiple hemangiomas

Exclusion Criteria:

* Patients older than 1 year of age.
* Patients with heart diseases.
* Patients with history of bronchspasm or wheezing.
* Patients with Hypotension.
* Patients with Hypertension.
* Premature infants with corrected age less than 5 weeks.
* Patients with conditions affecting blood glucose maintenance.
* Patients with liver failure.
* Patients with PHACES syndrome.

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete clinical clearance of hemangioma or reduction of hemangioma's volume. | within 9 months
  The efficacy of the treatment will be evaluated by complete clinical clearance of lesion (defined arbitrarily as >90% reduction in the size of Infantile Hemangioma as assessed by Physician Global Assessment) or after 9 months of treatment (primary end point) whichever is earlier for cutaneous infantile hemangiomas and by volume reduction of hemangiomas as evaluated by the proper imaging modalities ( Ultrasound, CT, or MRI) for non cutaneous hemangiomas.

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Teaching Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data is anticipated to become available on or after August 2022 and it will remain available for 5 years.
Access Criteria: will be provided later

REFERENCES:
- [Background] Darrow DH, Greene AK, Mancini AJ, Nopper AJ; SECTION ON DERMATOLOGY, SECTION ON OTOLARYNGOLOGY-HEAD AND NECK SURGERY, and SECTION ON PLASTIC SURGERY. Diagnosis and Management of Infantile Hemangioma. Pediatrics. 2015 Oct;136(4):e1060-104. doi: 10.1542/peds.2015-2485. PMID 26416931
- [Background] Darrow DH, Greene AK, Mancini AJ, Nopper AJ; SECTION ON DERMATOLOGY, SECTION ON OTOLARYNGOLOGY-HEAD & NECK SURGERY, AND SECTION ON PLASTIC SURGERY. Diagnosis and Management of Infantile Hemangioma: Executive Summary. Pediatrics. 2015 Oct;136(4):786-91. doi: 10.1542/peds.2015-2482. No abstract available. PMID 26416928
- [Background] Leaute-Labreze C, Harper JI, Hoeger PH. Infantile haemangioma. Lancet. 2017 Jul 1;390(10089):85-94. doi: 10.1016/S0140-6736(16)00645-0. Epub 2017 Jan 13. PMID 28089471
- [Background] HOLMDAHL K. Cutaneous hemangiomas in premature and mature infants. Acta Paediatr (Stockh). 1955 Jul;44(4):370-9. doi: 10.1111/j.1651-2227.1955.tb04151.x. No abstract available. PMID 13292246
- [Background] Amir J, Metzker A, Krikler R, Reisner SH. Strawberry hemangioma in preterm infants. Pediatr Dermatol. 1986 Sep;3(4):331-2. doi: 10.1111/j.1525-1470.1986.tb00535.x. PMID 3774653
- [Background] Hemangioma Investigator Group; Haggstrom AN, Drolet BA, Baselga E, Chamlin SL, Garzon MC, Horii KA, Lucky AW, Mancini AJ, Metry DW, Newell B, Nopper AJ, Frieden IJ. Prospective study of infantile hemangiomas: demographic, prenatal, and perinatal characteristics. J Pediatr. 2007 Mar;150(3):291-4. doi: 10.1016/j.jpeds.2006.12.003. PMID 17307549
- [Background] Margileth AM, Museles M. Cutaneous hemangiomas in children. Diagnosis and conservative management. JAMA. 1965 Nov 1;194(5):523-6. No abstract available. PMID 5897362
- [Background] Bennett ML, Fleischer AB Jr, Chamlin SL, Frieden IJ. Oral corticosteroid use is effective for cutaneous hemangiomas: an evidence-based evaluation. Arch Dermatol. 2001 Sep;137(9):1208-13. doi: 10.1001/archderm.137.9.1208. PMID 11559219
- [Background] Greenberger S, Boscolo E, Adini I, Mulliken JB, Bischoff J. Corticosteroid suppression of VEGF-A in infantile hemangioma-derived stem cells. N Engl J Med. 2010 Mar 18;362(11):1005-13. doi: 10.1056/NEJMoa0903036. PMID 20237346
- [Background] Crum R, Szabo S, Folkman J. A new class of steroids inhibits angiogenesis in the presence of heparin or a heparin fragment. Science. 1985 Dec 20;230(4732):1375-8. doi: 10.1126/science.2416056.
- [Background] Boon LM, MacDonald DM, Mulliken JB. Complications of systemic corticosteroid therapy for problematic hemangioma. Plast Reconstr Surg. 1999 Nov;104(6):1616-23. doi: 10.1097/00006534-199911000-00002. PMID 10541160
- [Background] Barlow CF, Priebe CJ, Mulliken JB, Barnes PD, Mac Donald D, Folkman J, Ezekowitz RA. Spastic diplegia as a complication of interferon Alfa-2a treatment of hemangiomas of infancy. J Pediatr. 1998 Mar;132(3 Pt 1):527-30. doi: 10.1016/s0022-3476(98)70034-4. PMID 9544915
- [Background] Deb G, Jenkner A, Donfrancesco A. Spastic diplegia and interferon. J Pediatr. 1999 Mar;134(3):382. doi: 10.1016/s0022-3476(99)70474-9. No abstract available. PMID 10064684
- [Background] Leaute-Labreze C, Dumas de la Roque E, Hubiche T, Boralevi F, Thambo JB, Taieb A. Propranolol for severe hemangiomas of infancy. N Engl J Med. 2008 Jun 12;358(24):2649-51. doi: 10.1056/NEJMc0708819. No abstract available. PMID 18550886
- [Background] Sans V, de la Roque ED, Berge J, Grenier N, Boralevi F, Mazereeuw-Hautier J, Lipsker D, Dupuis E, Ezzedine K, Vergnes P, Taieb A, Leaute-Labreze C. Propranolol for severe infantile hemangiomas: follow-up report. Pediatrics. 2009 Sep;124(3):e423-31. doi: 10.1542/peds.2008-3458. Epub 2009 Aug 10. PMID 19706583
- [Background] Buckmiller LM, Munson PD, Dyamenahalli U, Dai Y, Richter GT. Propranolol for infantile hemangiomas: early experience at a tertiary vascular anomalies center. Laryngoscope. 2010 Apr;120(4):676-81. doi: 10.1002/lary.20807. PMID 20112413
- [Background] Bagazgoitia L, Torrelo A, Gutierrez JC, Hernandez-Martin A, Luna P, Gutierrez M, Bano A, Tamariz A, Larralde M, Alvarez R, Pardo N, Baselga E. Propranolol for infantile hemangiomas. Pediatr Dermatol. 2011 Mar-Apr;28(2):108-14. doi: 10.1111/j.1525-1470.2011.01345.x. Epub 2011 Mar 8. PMID 21385205
- [Background] Cushing SL, Boucek RJ, Manning SC, Sidbury R, Perkins JA. Initial experience with a multidisciplinary strategy for initiation of propranolol therapy for infantile hemangiomas. Otolaryngol Head Neck Surg. 2011 Jan;144(1):78-84. doi: 10.1177/0194599810390445. PMID 21493392
- [Background] Holland KE, Frieden IJ, Frommelt PC, Mancini AJ, Wyatt D, Drolet BA. Hypoglycemia in children taking propranolol for the treatment of infantile hemangioma. Arch Dermatol. 2010 Jul;146(7):775-8. doi: 10.1001/archdermatol.2010.158. PMID 20644039
- [Background] Harrison DC, Meffin PJ, Winkle RA. Clinical pharmacokinetics of antiarrhythmic drugs. Prog Cardiovasc Dis. 1977 Nov-Dec;20(3):217-42. doi: 10.1016/0033-0620(77)90022-6. No abstract available. PMID 335439